CLINICAL TRIAL: NCT00387205
Title: An Open-Label, Phase Ib Study to Assess the Long Term Safety Profile of Pazopanib in Cancer Patients
Brief Title: Study To Assess Long Term Safety Of Pazopanib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: VEG105430; 2006-005528-17 (EudraCT Number)
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: chronic administration; monotherapy and combination therapies; solid; lapatinib (TYKERB, TYVERB); malignant tumor; Pazopanib; GW786034; cancer; safety
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Pazopanib monotherapy or in combination with lapatinib or other approved anti-cancer medications
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Pazopanib monotherapy or in combination with lapatinib or other approved anti-cancer medications

SUMMARY:
This study was a rollover study to evaluate the long term safety of pazopanib and to continue to provide pazopanib to patients who participated in a GSK sponsored pazopanib study until pazopanib is available commercially.

ELIGIBILITY:
Key Inclusion Criteria:

* Participated or completed a GSK sponsored pazopanib study and remains eligible for continued treatment with pazopanib and lapatinib (if on combination therapy).
* Able to understand and provide written informed consent
* Women and men agree to use protocol specific birth control measures

Key Exclusion Criteria:

* The subject has a treatment related serious adverse event that remains unresolved or unstable or had pazopanib permanently stopped in a previous study because of intolerate or because it was unsuccessful in treating your cancer
* If you are pregnant or breast feeding
* Your doctor does not think you would be a good candidate for the study
* Poorly controlled high blood pressure
* Subject is unwilling or unable to follow the procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2006-06-20 (Actual); Primary Completion 2013-02-13 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the long-term safety of repeat daily doses of pazopanib in cancer subjects with solid tumors | Subjects will stay on the study as long as they are benefiting from treatment, have not met one of the stopping criteria, or experienced a toxicity up to 72 months.
  To evaluate the safety assessments; adverse events, vital signs, physical examinations, electrocardiograms, multi-gated acquisition scans or echocardiograms (only for patients on pazopanib and lapatinib combination therapy), and clinical laboratory assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- United States (15):
  - Novartis Investigative Site, Duarte, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Tacoma, Washington
- Novartis Investigative Site, Lyon, France
- Novartis Investigative Site, Singapore, Singapore
- United Kingdom (2):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No